CLINICAL TRIAL: NCT03884088
Title: Comparison of Sensitivity of the Subjective Balance Tests
Brief Title: Comparison of Subjective Balance Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GO 19/29
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Balance; Posture
Keywords: Balance; Limits of Stability; Postural Sway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Balance analysis (Experimental): Balance will be assessed by Computerized Balance system and subjective balance tests.
  Interventions: Other: Limits of Stability
- Control Group: Balance analysis (Active Comparator): Balance will be assessed by Computerized Balance system and subjective balance tests.
  Interventions: Other: Limits of Stability

INTERVENTIONS:
Other: Limits of Stability — Balance analysis is assessment method to estimate fall of risk and deterioration of postural control.
  Other Names: Postural Sway test; Berg Balance Scale; Y Balance Test; Romberg Balance Test; One-Leg Stance Test; Tinetti Balance Test; Timed up an go test; Functional Reach Test

SUMMARY:
There is many subjective balance tests to evaluate static and dynamic balance. But, there is no sufficient information about which balance test is the most sensitive test to evaluate balance. Therefore, the aim of this study is to compare of sensitivity of the subjective balance tests with an objective system.

DETAILED DESCRIPTION:
In the clinical setting, many balance tests are used for evaluating balance in individuals. These tests are utilized to assess both static and dynamic balance. However, sufficient research has not been conducted to decide which subjective balance test is more sensitive than the other tests. Therefore, the aim of this study is to compare of sensitivity of the subjective balance tests with an objective system.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years,
* To be a volunteer to participate

Exclusion Criteria:

* orthopedic problems affecting gait and stance
* visual, auditory, orientational problems that could affect study results,
* Walking with assist device
* Having a neurological disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Limits of Stability | 15 minutes
  Limits of stability test evaluates dynamic balance of participants. Computerized balance system measured limits of stability for forward, backward, right and left side movements. It calculates the maximum distance a person can lean without losing balance. The unit of measure is centimeters. The higher value is indicated the better balance
Postural Sway | 15 minutes
  Postural sway in centimeters by computerized balance system

SECONDARY OUTCOMES:
Timed up and go test | 15 minutes
  Timed up and go test evaluates dynamic balance of participants. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.Timed up and go test measure is second. The lower values indicates the better balance
Functional reach test | 15 minutes
  Functional reach test evaluates dynamic balance by measuring the limits while the patient reaches forwards as far as possible. The test measure is centimeters. A higher score indicates better dynamic balance.
One-leg stance test | 15 minutes
  One-leg stance test evaluates static balance of the participants. Participants would ask to maintain their static balance by standing one-lag stance. The test measure is second. A higher score indicated better static balance
Romberg test | 15 minutes
  Romberg test is used to evaluate static balance. Participants would ask to maintain their balance with their feet together (touching each other). The test measure is second. Higher score indicated better balance.
Berg balance scale | 15 minutes
  Berg balance scale is used for functional balance. participants are asked to perform 14 tasks frequently used in daily life activities. The highest possible score is 56 points. A higher score indicates better balance.
Balance scale | 15 minutes
  Balance scale which is developed by Tinetti is used to evaluate functional balance. This test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totalling 28. The lower the score on the scale, the higher the risk of falling.
Y balance test | 15 minutes
  Y balance test is used to evaluate dynamic balance. The Y balance test has the patient stand on one leg while reaching out in 3 different directions with the other lower extremity. They are anterior, posteromedial and posterolateral. The test measures in centimeters. The higher score indicates better balance

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No